CLINICAL TRIAL: NCT04122365
Title: Effectiveness of Chest Wall Mobilization Program in Improving Respiratory Function for Patients With Chronic Obstructive Pulmonary Disease. A Randomized Controlled Trial
Brief Title: Effectiveness of Chest Wall Mobilization Program in Improving Respiratory Function for Patients With COPD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: COPD Study
Record Dates: First submitted 2019-07-23; First posted 2019-10-10 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2019-05

CONDITIONS: COPD
Keywords: Chest Wall Mobilization Program; Respiratory Function
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Respiratory Aspiration

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional group (Experimental): Chest Wall Mobilization Program
  Interventions: Other: Chest Wall Mobilization Program
- Control Group (Other): Routine limbs exercises and education
  Interventions: Other: Control

INTERVENTIONS:
Other: Chest Wall Mobilization Program — Soft tissue therapy and joints mobilization
  Arms: Interventional group
Other: Control — Routine limbs exercises and education
  Arms: Control Group

SUMMARY:
Patients with severe COPD will be recruited from the Respiratory Outpatient Clinic of Kowloon Hospital.

Baseline (pre-intervention) assessment for all recruited subjects will be conducted by one physiotherapist assessor who is blinded to the group allocation of the subject for respiratory function, musculoskeletal performance, physical performance and quality of life. Then, the subjects will be randomly allocated into either the intervention group with therapist-assisted chest wall mobilization exercises, low intensity walking exercise, home exercises and education sessions or the control group with low intensity walking exercise, home exercises and education sessions. The intervention program will last for 6 weeks with 2 sessions / week (i.e. a total of 12 sessions) in accordance to the recommendation for exercise training programs for patients with COPD by the American College of Sports Medicine. Post-program evaluation will be conducted upon program completion at 6 week.

A follow-up session on 3 month after the completion of the program will be carried out to evaluate the cumulative effect of the chest wall mobilization program on respiratory function, musculoskeletal performance, exercise performance and quality of life of the patients.

DETAILED DESCRIPTION:
I. Intervention for Study Group

Structured Chest Wall Mobilization Program

Chest Wall Mobilization Chest wall mobilization is one of the important techniques in chest physical therapy for increasing chest wall mobility and improving ventilation. Either passive or active chest mobilizations help to increase chest wall mobility, flexibility, and thoracic compliance. The mechanism of this technique increases the length of the intercostal muscles and therefore helps in performing effective muscle contraction. It improves the biomechanics of chest movement by enhancing direction of anterior-upward movement of lower costal and downward movement of diaphragm. Maximal relaxed recoiling of the chest wall helps in achieving effective contraction of intercostal muscle. Chest wall mobilization with breathing exercise was showed to effect clinical benefit in chronic lung disease especially COPD with lung hyperinflation or barrel-shaped chest. The technique of chest wall mobilization helps in chest wall flexibility, respiratory muscle function and ventilatory pumping, which helps to reduce dyspnoea and respiratory accessory muscle use.

The chest wall mobilization techniques include:

1. Lateral flexion of chest wall
2. Chest wall extension
3. Lateral gliding of thoracic spine
4. Pectoralis major muscle stretching

There is no standard of practice found on the current studied chest wall mobilization. As good practice for quality and safety assurance, the studied program was evaluated by two independent Physiotherapists expert with post-graduate qualification in Manual Therapy recognised by Physiotherapists Board of Hong Kong Government and the International Federation of Orthopaedic Manipulative Physical Therapists of World Confederation of Physical Therapy. Chest wall mobilization will be performed in a therapist-assisted manner by a single trained and certified American College of Sports Medicine (ACSM) Clinical Exercise Physiologist with more than 10 years' experience working in the speciality with chronic respiratory patients in respiratory medicine.

Subjects will be placed in the sitting position, lying on the back or sidelying position with knees bent to correct the lumbar curve, repositioning of the scapular waist as well as scapular and arm abduction in order to prevent postural compensations. Stretching was performed bilaterally as follows:

1. Lateral flexion of chest wall Patient in supine and lateral position on a foam roller in the infra-axillary region, forearms flexed and hands resting on the occipital region; the therapist used both palmar region hand's to mobilize the ribs in the cranial and caudal direction.
2. Chest wall extension Patient in supine lying on a foam roller in the mid-thoracic region, raise the arm over the head and grasp hold on a fixed wall bar about 10 inches from the surface of the plinth.
3. Lateral gliding of thoracic spine It is a non-thrust transverse vertebral pressure as described by Maitland et al 2005. Patients in prone lying, arms to the side and head in a 'forehead rest position'. Mobilization was applied to the whole thoracic spine. The spinous process of T1 was identified by first locating C6 using the cervical extension method and then counting caudally. The therapist stood at the level of the vertebra to be mobilized on one side of the subject. The pad of the therapist's non-dominant thumb was placed in contact with the lateral aspect of the spinous process of T1, whereas the dominant thumb was placed on the dorsal side of the other thumb. Pressure was applied to the spinous process to produce small amplitude, low velocity oscillations into resistance to the end-range of the vertebra (Grades IV). This procedure was performed for 30 seconds, and then sequentially applied to the next caudal level. The same pattern of application was used on the patient's contralateral side.
4. Pectoralis major stretching Patient in supine position, on the side to be stretched, the patient´s arm was abducted, forearm flexed and hand resting on the occipital region. The displacement was performed with one of the therapist's hands on the upper third of the arm and the other on the lateral region of the upper chest, following the direction of muscle fibres.

The therapist-assisted chest wall mobilization for stretching follow the guidelines of general stretching for skeletal muscles. Static stretching will be performed with the therapist assisted the movement to the available range and hold in that position with the muscle on tension to a point of a stretching sensation. The stretching will be carried out during the expiratory phase with two sets of ten consecutive incursions for each position and a one-minute rest between the series. The holding of the stretching sensation should last for 10 seconds. The intervention will be around 20 minutes in total.

For the participants in the Control group, they will be asked to stay in supine, sidelying and prone positions for around 20 minutes to standardize the treatment time and effect of positioning.

Intervention Group Home Exercise Program For maintenance of the intervention effect and further improvement of chest wall mobility as well as soft tissues elasticity. Self-stretching exercises of trunk extension, rotation, side flexion as well as stretching of the pectoralis major muscle will be taught to the patients as home exercise program. Participants will be asked to perform the home exercise program for 15 minutes, 3 days /week for 6 weeks. An individual exercise log-book with the diagram of the stretching exercises will be given to the subjects to follow the exercises and record down their participation. Weekly telephone contact to participant will be given for motivation and encouragement of program adherence and completing the log books.

II. Intervention for Control Group Subjects in the control group will be asked to maintain their physical activity level as usual. A 15-minute simple stretching exercise on large muscle group will be taught for standardization as a home exercise program. Five stretching exercises for arms and legs will be taught to the patient as a home exercise program. Participants will be asked to perform the home exercise program for 15 minutes, 3 days /week for 6 weeks. An individual exercise log-book with the diagram of the stretching exercises will be given to the subjects to follow the exercises and record down their participation. Same weekly telephone contact to participant will be given for motivation and encouragement of program adherence and completing the log books as that in intervention group.

III. Common Program for Both Groups Standardized Walking Exercise Exercise will be performed on a Gaitkeeper Mobility Research 2000T electronic treadmill (Cortland, New York) set at zero inclination during subject's follow-up visit at Physiotherapy Department of Kowloon Hospital. Each participant will perform 15 minutes supervised walking exercise at a speed maintain with the participant's target heart rate zone of 60-80% Heart Rate Maximum for cardiovascular training. Besides, the oxygen saturation during walking will be kept above 88%. An oximeter will be used to adjust walking speed and monitoring of HR and oxygen saturation.

Standardized Educational Session Three educational sessions (30 minutes for each session) will be included for both intervention group and control group at Physiotherapy Department of Kowloon Hospital. The content of the education include self-management of bronchial hygiene, breathing re-training, relaxation techniques and the importance of exercise. Education pamphlets will be given to both groups of patients.

ELIGIBILITY:
Inclusion Criteria:

1. COPD patients in out-patient setting: Patients with FEV1/FVC < 0.70 and

GOLD stage III ( Severe) :

30% < or = FEV1 < 50% predicted

*GOLD - Global Initiative for Chronic Obstructive Lung Disease

2. Ambulatory

3. Able to communicate

4. Competent to give written consent

Exclusion Criteria:

1. Contraindications to chest wall mobilization:

   * Severe and unstable rib fracture
   * Metastasis bone cancer
   * Tuberculosis spondylitis
   * Severe osteoporosis
2. Hospitalization due to acute exacerbation of COPD in recent 1 month
3. Current Smoker

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-10 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Lung Function | 4.5 months
  FEV1, FVC and Ratio
Respiratory Muscles Function | 4.5 months
  Maximum Inspiratory Pressure, Maximum Expiratory Pressure

SECONDARY OUTCOMES:
Cervical and Thoracic Range of Movement | 4.5 months
  Measurement of cervical and thoracic range of movement with motion sensor in degree
Cervical and Respiratory Muscles Activity | 4.5 months
  Electromyography measurement of cervical and respiratory muscles
Respiratory Muscle Oxygenation | 4.5 months
  Near Infrared Spectroscopy on intercostal muscles
Thoracic Excursion | 4.5 months
  Measurement of upper and lower thoracic expansion using tape measure in cm
Six-Minute Walk Test | 4.5 months
  Measurement of distance, SpO2, Heart rate
Pressure Pain Threshold | 4.5 months
  Use Pressure algometer for measure the pressure pain threshold
Visual Analogue Scale | 4.5 months
  A 10cm line to rate his or her pain.
St George's Respiratory Questionnaire | 4.5 months
  3 Domains: Symptoms, Activity and Impacts. A total score 0-100.

CONTACTS AND LOCATIONS:
Overall Officials: TSUI, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- Kowloon Hospital, Kowloon, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Balady, G.J., Berra, K.A., Golding, L.A., Gordan, N.F., Mahler, D,A., Myers, J.N., & Sheldahl, L.M. (2017). ACSM's Guidelines for Exercise Testing and Prescription. Philadelphia: Lippincott Williams & Wilkins.
- [Background] de Sa RB, Pessoa MF, Cavalcanti AGL, Campos SL, Amorim C, Dornelas de Andrade A. Immediate effects of respiratory muscle stretching on chest wall kinematics and electromyography in COPD patients. Respir Physiol Neurobiol. 2017 Aug;242:1-7. doi: 10.1016/j.resp.2017.03.002. Epub 2017 Mar 10. PMID 28286249
- [Background] Duiverman ML, de Boer EW, van Eykern LA, de Greef MH, Jansen DF, Wempe JB, Kerstjens HA, Wijkstra PJ. Respiratory muscle activity and dyspnea during exercise in chronic obstructive pulmonary disease. Respir Physiol Neurobiol. 2009 Jun 30;167(2):195-200. doi: 10.1016/j.resp.2009.04.018. Epub 2009 May 3. PMID 19406254
- [Background] Ekstrum, J.A., Lisa L. Black & Karen A. Paschal (2009). Effects of a Thoracic Mobility and Respiratory Exercise Program on Pulmonary Function and Functional Capacity in Older Adults. Physical & Occupational Therapy in Geriatrics, 27(4), 310-327.
- [Background] Engel RM, Vemulpad SR, Beath K. Short-term effects of a course of manual therapy and exercise in people with moderate chronic obstructive pulmonary disease: a preliminary clinical trial. J Manipulative Physiol Ther. 2013 Oct;36(8):490-6. doi: 10.1016/j.jmpt.2013.05.028. Epub 2013 Sep 17. PMID 24053900
- [Background] Engel RM, Vemulpad S. The effect of combining manual therapy with exercise on the respiratory function of normal individuals: a randomized control trial. J Manipulative Physiol Ther. 2007 Sep;30(7):509-13. doi: 10.1016/j.jmpt.2007.07.006. PMID 17870419
- [Background] Engel R, Vemulpad S. The role of spinal manipulation, soft-tissue therapy, and exercise in chronic obstructive pulmonary disease: a review of the literature and proposal of an anatomical explanation. J Altern Complement Med. 2011 Sep;17(9):797-801. doi: 10.1089/acm.2010.0517. Epub 2011 Aug 12. PMID 21838523
- [Background] Gosling, C., & Williams, K.A. (2004). Comparison of the effects of thoracic manipulation and rib raising on lung function of asymptomatic individuals. Journal of Osteopathic Medicine, 7, 103.
- [Background] Heneghan NR, Adab P, Balanos GM, Jordan RE. Manual therapy for chronic obstructive airways disease: a systematic review of current evidence. Man Ther. 2012 Dec;17(6):507-18. doi: 10.1016/j.math.2012.05.004. Epub 2012 Jun 15. PMID 22703901
- [Background] Heneghan, N., Adab, P., Jackman, S., & Balanos, G. (2015). Musculoskeletal dysfunction in chronic obstructive pulmonary disease (COPD): An observational study. International Journal of Therapy and Rehabilitation, 22(3), 119-128.
- [Background] Kaneko H, Shiranita S, Horie J, Hayashi S. Reduced Chest and Abdominal Wall Mobility and Their Relationship to Lung Function, Respiratory Muscle Strength, and Exercise Tolerance in Subjects With COPD. Respir Care. 2016 Nov;61(11):1472-1480. doi: 10.4187/respcare.04742. Epub 2016 Oct 18. PMID 27794081
- [Background] Kelzuyuki, Tabira, Sekikawa, Noriko, Iwashiro, Motoki, Kawato, Seiji, Sekikawa, Kiyokazu, Kawamata, Mikio, Oike, Takayuki. (2007). The immediate effect of chest mobilization tech. in patients of COPD. The Journal of Japanese Physical Therapy Association, 34(2), 59-64.
- [Background] Leelarungrayub D, Pothongsunun P, Yankai A, Pratanaphon S. Acute clinical benefits of chest wall-stretching exercise on expired tidal volume, dyspnea and chest expansion in a patient with chronic obstructive pulmonary disease: a single case study. J Bodyw Mov Ther. 2009 Oct;13(4):338-43. doi: 10.1016/j.jbmt.2008.11.004. Epub 2009 Jan 29. PMID 19761957
- [Background] Parmar, D., & Bhise, A. (2015). The immediate effect of Chest mobilization technique on chest expansion in patients of COPD with restrictive impairment. International Journal of Science and Research, 4(6), 2413-2416.
- [Background] Putt MT, Watson M, Seale H, Paratz JD. Muscle stretching technique increases vital capacity and range of motion in patients with chronic obstructive pulmonary disease. Arch Phys Med Rehabil. 2008 Jun;89(6):1103-7. doi: 10.1016/j.apmr.2007.11.033. PMID 18503806